CLINICAL TRIAL: NCT00259259
Title: The Effect of Functional Lipids on Appetite Regulation in Man
Brief Title: Functional Lipids and Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danisco (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: (KF) 01 275625; B218
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-09

CONDITIONS: Obesity
Keywords: Appetite regulation; Hormones; Energy intake
MeSH Terms: conditions — Obesity | interventions — salatrim

INTERVENTIONS:
Behavioral: SALATRIM

SUMMARY:
To evaluate the short-term effects of structured lipids on appetite regulation.

DETAILED DESCRIPTION:
Background Obesity is a major health problem worldwide, and it is a risk factor for several chronic disorders. Even small changes in energy intake, leading to a positive balance may lead to weight gain over time. Thus, slight modifications in food intake, such as the inclusion of foods that effect energy balance, may prevent weight gain and even facilitate weight loss. Replacing dietary fat with low-calorie fat (LCF), such as modified triglycerides with medium and long chained PUFA.may be an efficient way to reduce body fat.

Bray et al. (2002) has shown a sustained weight loss of ~6 kg over a 9 month period where one-third of a fat-reduced diet (25% fat) was replaced by olestra. This weight loss can not solely be explained by the decreased caloric content of olestra. Thus, inhibition of appetite leading to lower food intake, may be a potential mechanism of the observed weight loss.

A reduced absorption of LCF leaves undigested fatty acids in the middle and lower intestine, which may generate increased feelings of satiety and decrease caloric intake due to regulating peptides and hormones such (CCK, GLP-1, etc.). In addition, intraduodenal fatty acids may also promote distension of the stomach and distension of the intestine, which are well-known gastrointestinal signals controlling mechanisms for food intake.

Taken together, in addition to the acute reduction in caloric intake, LCF may encourage a gastrointestinal hormone response promoting beneficial effects on appetite regulation and energy balance.

Aims To evaluate the short-term effects of LCF on

Primary:

* Appetite sensations after a meal (VAS)
* Postprandiel secretion of appetite regulating hormones
* Ad libitum caloric intake 4,5-h subsequent to a fixed meal

Secondary:

• Palatability of the test meal

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* Normal weigh, e.i. BMI between 18,5-25 kg/m2
* age 18-40 years

Exclusion Criteria:

* donation of blood 3 monhts prior or during the study
* gastrointestinal disorders, diabetes, hypertension, hyperlipidemia, chronic infectious disease
* smoking
* consumption of more than 21 alcoholic drinks/week
* elite athletes
* on mediation
* diet supplements

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2005-10; Study Completion 2005-12

PRIMARY OUTCOMES:
Appetite
energy intake
Hormones

SECONDARY OUTCOMES:
Palability

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Proffessor, Principal Investigator — Department of human nutrition, The Royal Veterinary and Agricultural University
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg C, Copenhagen, Denmark